CLINICAL TRIAL: NCT06481553
Title: Real-world Study of the Efficacy and Safety of Paclitaxel Liposome Combined With Anti-HER-2 Monoclonal Antibody as First-line Salvage Treatment of HER-2 Positive Advanced Breast Cancer
Brief Title: RWS of Paclitaxel Liposome Combined With Anti-HER-2 Monoclonal Antibody
Status: Active, not recruiting | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 24/103-4383
Record Dates: First submitted 2024-06-25; First posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer Stage IV
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: first line treatment — Paclitaxel liposome in combination with trastuzumab (or trastuzumab biosimilar, or pyrotinib) ± pertuzumab ± other chemotherapy drugs (such as capecitabine, carboplatin, gemcitabine) may be used for HER-2 positive patients, with the addition of endocrine therapy for triple-positive patients.

SUMMARY:
This is a retrospective, single-arm real-world study based on the National Anticancer Drug Clinical Application Monitoring Network database.The aim of this study is to evaluate the efficacy and safety of paclitaxel liposome combined with anti-HER-2 monoclonal antibody as first-line salvage treatment for HER-2 positive advanced breast cancer. It seeks to understand the application patterns, efficacy, and safety of paclitaxel liposome combined with anti-HER-2 monoclonal antibody in real-world settings, providing patients with safer treatment options.

DETAILED DESCRIPTION:
The National Anticancer Therapy Data Surveillance System (NATDSS) is the largest oncology diagnosis and treatment database in China to date, covering patient data from over 1400 oncology hospitals and integrated hospitals. It has collected data from approximately 15 million cancer patients since 2013, including mortality information obtained from the CDC death registration database.

Paclitaxel liposome was introduced to the market in 2004 as a formulation of paclitaxel. It utilizes nanotechnology to encapsulate the poorly water-soluble paclitaxel within a lipid bilayer of liposomes, solving the issue of paclitaxel& low solubility in water. Paclitaxel liposome no longer employs polyoxyethylated castor oil as a solvent. While ensuring efficacy, it reduces the risk of associated adverse drug reactions (such as severe allergic reactions), thereby enhancing the tolerance of cancer patients.

Although paclitaxel liposome is widely used in HER-2 positive advanced breast cancer, there is currently no research on the efficacy and safety of combining paclitaxel liposome with anti-HER-2 monoclonal antibodies as first-line salvage treatment of HER-2 positive advanced breast cancer.

This study aims to conduct a real-world study on the efficacy and safety of combining paclitaxel liposome with anti-HER-2 monoclonal antibodies as first-line salvage treatment of HER-2 positive advanced breast cancer based on the NATDSS

ELIGIBILITY:
inclusion criteria:

1. Patients with unresectable or metastatic HER-2 positive breast cancer (immunohistochemistry 3+ or FISH positive) have received at least 2 cycles of salvage treatment with paclitaxel liposome in combination with anti-HER-2 therapy (monotherapy or dual-targeted therapy) ± other chemotherapy drugs (such as capecitabine, carboplatin, gemcitabine) as first-line treatment.
2. Patients with no visceral metastases, but only have bone metastases or multiple lymph node metastases are eligible for inclusion.
3. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2. Expected survival of at least 3 months.

exclusion criteria：

1. Accompanied by other secondary malignant tumors.
2. Male breast cancer or bilateral breast cancer.
3. brain metastasis

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with unresectable or metastatic HER-2 positive breast cancer (immunohistochemistry 3+ or FISH positive) have received at least 2 cycles of salvage treatment with paclitaxel liposome in combination with anti-HER-2 therapy (monotherapy or dual-targeted therapy) ± other chemotherapy drugs (such as capecitabine, carboplatin, gemcitabine) as first-line treatment.
Sampling Method: Non-Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | 5-year
  The time from the initiation of drug treatment until death due to any cause
real world progress free survival（rwPFS） | 5-year
  The time from the initiation of drug treatment until disease progression (as evaluated by medical records or imaging records) or death, whichever comes first, can be considered as the time to event endpoint in the study. This endpoint can be represented as the time to treatment change in case PFS data is missing.

SECONDARY OUTCOMES:
Time To Progression | 5-year
  The time from the initiation of drug treatment until disease progression (as evaluated by medical records or imaging records)，Excluding death
Time to Treatment Failure | 5-year
  The time from the initiation of drug treatment until termination of treatment for any reason (including disease progression, unacceptable toxicity, and death)

CONTACTS AND LOCATIONS:
Overall Officials: Zhou G Hui, MD, Study Chair — National Cancer Center/Cancer Hospital
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: No